CLINICAL TRIAL: NCT03902626
Title: Understanding Attitudes and Beliefs of Undergraduate Medical and Physiotherapy Students - a Longitudinal Study
Brief Title: Chronic Pain Attitudes Medical and Physiotherapy Students
Status: Completed | Type: Observational
Sponsor: Teesside University (Other)
Collaborators: Glasgow Caledonian University (Other); University of Glasgow (Other)
Responsible Party: Principal Investigator, Mrs Jagjit Mankelow, Principal investigator, Teesside University
Other Study IDs: 062/18
Record Dates: First submitted 2019-04-02; First posted 2019-04-04 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Chronic Low Back Pain
Keywords: attitudes; chronic low back pain; functionality; healthcare professional students
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Physiotherapy students: Degree course
  Interventions: Other: Physiotherapy students
- Medical students: Degree course
  Interventions: Other: Medical students

INTERVENTIONS:
Other: Physiotherapy students
  Groups: Physiotherapy students
Other: Medical students
  Groups: Medical students

SUMMARY:
This is an analysis of data collected from 2009-2014 from medical students at GCU and physiotherapy students at UoG measuring attitudes towards patients with chronic low back pain and their functionality.

DETAILED DESCRIPTION:
This is longitudinal study with the data collected from 2009-2014 from medical students and physiotherapy students at two different Scottish universities measuring attitudes towards patients with chronic low back pain and their functionality. The outcome measure used was HC-PAIRS the original 15 point Likert Scale. Data was analysed using SPSS (version 25). All data was found to be normally distributed. Descriptive statistics were presented as mean (Standard Deviation). Inferential statistics were carried out using a two-way ANOVA with year of study and discipline of degree as independent variables with post hoc analysis. A p-value of <0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

-Engaged in the 2009 physiotherapy degree at Two Scottish universities

Exclusion Criteria:

-Anyone who is not on the above degree courses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Students registered for the 2009 physiotherapy and medical degree at two Scottish universities
Sampling Method: Non-Probability Sample
Enrollment: 267 (Actual)
Dates: Start 2009-09-01 (Actual); Primary Completion 2013-01-01 (Actual); Study Completion 2013-01-01 (Actual)

PRIMARY OUTCOMES:
HC-PAIRS (Health care providers pain and impairment relationship scale) | 1 x year for duration of degree course at start of first semester
  15 point Likert Scale ranging in score from 15 to105 with a low score reflecting an attitude towards patients with pain and their functionality which is in keeping with best evidence research and scientific knowledge. Subscales are not valid for this outcome measure.